CLINICAL TRIAL: NCT06092476
Title: A Randomized Double-blind Sham-controlled Trial to Evaluate Efficacy+Safety of Revita Duodenal Mucosal Resurfacing (DMR) Treatment Paradigm+Retreatment in Patients With Type 2 Diabetes Using Non-insulin Glucose Lowering Medications (REMIND)
Brief Title: Trial to Evaluate Efficacy+Safety of Revita DMR Treatment Paradigm 1 and Retreatment in Type 2 Diabetes Patients
Acronym: REMIND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Fractyl Health Inc. (Industry)
Responsible Party: Principal Investigator, Jacques J.G.H.M. Bergman, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL82963.018.23
Record Dates: First submitted 2023-09-22; First posted 2023-10-23 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Duodenal ablation; Endoscopy; Duodenal Mucosal Resurfacing
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The study is a single-center, randomized, double-blind, sham-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, both the study team and the study subjects are blinded to the treatment through the 24 week follow-up visit. While the endoscopist is not blinded to individual treatments, he is blinded to cohort level data and is not responsible for patient follow-up. At the 24 week visit, the subject and study team are unblinded. The subjects who received the sham treatment undergo DMR treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- DMR procedure (Active Comparator): Patients receive Revita® DMR Treatment Paradigm 1. After unblinding at 24 weeks, they receive retreatment.
  Interventions: Device: Revita® DMR Treatment
- Sham procedure (Sham Comparator): Patients receive a sham procedure. After unblinding takes place at 24 weeks, patients receive a Revita® DMR Treatment Paradigm 1. 48 weeks after initial sham (= 24 weeks after first DMR) patients may receive retreatment, if they want to.
  Interventions: Other: Sham procedure

INTERVENTIONS:
Device: Revita® DMR Treatment — The Revita® System is an endoscopic treatment consisting of a single catheter and console designed to lift the duodenal mucosa with saline followed by controlled circumferential hydrothermal ablation of the mucosa. For this study Revita® DMR procedure will be conducted as follows:
  DMR Treatment Paradigm 1- After initial 2 Lift and Ablate step, remaining Lift: Ablate steps will be conducted in 1:1 manner.
  Other Names: Revita® DMR Treatment Paradigm 1; Revita Duodenal Mucosal Resurfacing
  Arms: DMR procedure
Other: Sham procedure — The sham control for the Revita DMR procedure.
  Arms: Sham procedure

SUMMARY:
The objective of this study is to evaluate feasibility, safety, and efficacy of endoscopic DMR Treatment Paradigm 1 (compared to sham) and to evaluate feasibility, safety, and efficacy of re-treatment with DMR at 24 weeks (compared to baseline and a single DMR procedure) in patients with type 2 diabetes with non-insulin glucose lowering medications.

DETAILED DESCRIPTION:
The objective of this study is to evaluate feasibility, safety, and efficacy of endoscopic DMR Treatment Paradigm 1 (compared to sham) and to evaluate feasibility, safety, and efficacy of re-treatment with DMR at 24 weeks (compared to baseline and a single DMR procedure) in patients with type 2 diabetes with non-insulin glucose lowering medications.

The aimed effect is an adequate or improved glucose regulation and a decrease of HbA1c. Secondary effects include improved cardiovascular, hepatic, and metabolic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with Type 2 Diabetes.
2. Age ≥ 18 to ≤ 75 years.
3. Insulin naïve patients who are on stable dose (maximally approved or tolerated dose) of 2 or more glucose lowering drugs, including metformin, sulphonylurea (SU), (sodium-glucose cotransporter-2) inhibitors (SGLT-2i), Glucagon-like peptide-1 receptor agonists (GLP-1RA) or dipeptidyl peptidase 4 inhibitor (DPP-4i) and/or, thiazolidinedionderivaten (TZD) for at least 12 weeks.
4. BMI ≥ 24 and ≤ 40 kg/m2
5. HbA1c of ≥ 54 mmol/mol (7.5%) and ≤ 86 mmol/mol (10.0%).
6. Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation.

Exclusion Criteria:

1. Uncontrolled hyperglycemia with a glucose level >270 mg/dl (>15.0 mmol/L) after an overnight 8-hour fasting at the end of run-in and confirmed by a second measurement on the consecutive day.
2. Subjects who are using insuline.
3. Known case of absolute insulin deficiency as indicated by a fasting plasma C-peptide value of <0.6 ng/ml (<0,2 nmol/L).
4. Diagnosis of autoimmune diabetes/Type 1 diabetes mellitus, monogenic (neonatal or maturity onset diabetes of the young (MODY)) diabetes or Type 1 diabetes in adults/latent autoimmune diabetes of adults (LADA).
5. History of more than 1 severe hypoglycemia episode or unawareness within past 6 months in which third party assistance was needed.
6. Clinically significant valvular heart disease or severe aortic stenosis.
7. Acute coronary syndrome (non-ST wave elevated myocardial infarction (STEMI), STEMI and unstable angina pectoris), stroke or transient ischemic attack within the past 3 months.
8. Indication of acute liver disease, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN).
9. Presence of acute or chronic active hepatitis B or C (except if hepatitis C is cured) or cirrhosis; or hepatic decompensation during the last 6 months; or alcoholic or autoimmune chronic hepatitis.
10. Impaired renal function, defined as estimated Glomerular Filtration rate (eGFR) < 45 ml/min/1.73m2 or end stage renal failure or on dialysis.
11. Diagnosed with esophageal motility disorder or Glomerular Filtration rate (GERD) gr 3 or diagnosed during screening endoscopy.
12. Known history of a structural or functional disorder of the stomach, e.g. active gastric ulcer, chronic gastritis, gastric varices, hiatal hernia, stomach cancer or any other disorder of the stomach.
13. Previous GI surgery that could affect the ability to treat the duodenum such as patients who have had a Billroth 2, Roux-and-Y gastric bypass, gastric sleeve or other similar procedures.
14. Known intestinal autoimmune disease, including Celiac disease, or pre-existing symptoms of lupus erythematosus, scleroderma, or other autoimmune connective tissue disorder, which affects the small intestine.
15. Patients with active helicobacter pylori infection. Patients may be enrolled if they had history of h-pylori infection and were successfully treated.
16. History of active malignancy or partial remission from clinically significant malignancy within the past 5 years. With the exception of basal or squamous cell skin cancer or carcinoma in situ or those received curative treatment and in complete remission for 5 years or if subject confirmed as cancer free.
17. Blood dyscrasias or any disorders causing hemolysis or unstable Red Blood Cells (sickle cell trait is allowed).
18. Known case of severe peripheral vascular disease.
19. Clinically active systemic infection.
20. Known immunocompromised status, including individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months, clinically significant leukopenia or positive for the human immunodeficiency virus (HIV), on potential immunosuppressants.
21. Current treatment with systemic steroids or change in dosage of thyroid hormones within 6 weeks prior to consent or any other uncontrolled endocrine disorder.
22. Use of anticoagulation therapy (such as warfarin, coumadin, Novel Oral AntiCoagulants (NOAC) or anti-platelet agents (such as thienopyridine) which cannot be discontinued for 5-7 days or 2 drug half-lives before the procedure; Acetylsalicylic acid does not need to be discontinued.
23. Actively participating in weight loss program or using medications for weight loss 3 months prior to randomization.
24. General contraindications to deep or conscious sedation or general anesthesia or high risk (e.g., American Society of Anesthesiologists Classification (ASA) 4 or higher) or contraindications to upper GI Endoscopy.
25. Nursing or Pregnant women or women of child bearing potential who are unwilling to practice acceptable method of birth control.
26. History of alcohol, legal or illegal drug and substance abuse.
27. Intake of an investigational drug in another trial within 30 days prior to consent or active participation in another clinical trial of an investigational drug or device.
28. Any other clinical or mental condition which would jeopardize subject's safety or makes subject a poor candidate for clinical trial participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint | 12 weeks post DMR and 12 weeks post retreatment with DMR
  Safety endpoint is evaluated 12 weeks post DMR and 12 weeks post retreatment with DMR
  - Number (percentage) of patients experienced device and procedure-related Serious Adverse Events (SAEs), Unanticipated Device Effects (UADEs), Serious Adverse Device Effects (SADEs), Suspected Unexpected Serious Adverse Reaction (SUSARs)
Feasibility endpoint 1 | During procedure
  Feasibility endpoint is evaluated during and after the procedure:
  - Number of ablations, whether a DMR was successful (>3 ablations)
Feasibility endpoint 2 | During procedure
  Feasibility endpoint is evaluated during and after the procedure:
  - Procedure time, defined as time between catheter in and catheter out.
Efficacy endpoint 1 | 24 weeks post DMR/sham
  Efficacy is evaluated at 24 weeks compared to baseline and sham:
  - Mean change in Fasting Plasma Glucose (FPG)/Flash Glucose Monitoring (FGM)
Efficacy endpoint 2 | 24 weeks post DMR/sham
  Efficacy is evaluated at 24 weeks compared to baseline and sham:
  - Change in HbA1c

SECONDARY OUTCOMES:
Secondary safety endpoint | Through study completion, an average of 1 or 1,5 years
  Secondary safety endpoint is evaluated during follow-up and compared to baseline and sham at week 24 and compared to baseline and 12 weeks after (re)-DMR for all patients: incidences and event rates of hypoglycemic events during complete study period
Efficacy endpoint 1: mean change in HbA1c | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 1: mean change in HbA1c
Efficacy endpoint 2: mean Change in Fasting Glucose | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 2: mean Change in Fasting Glucose
Efficacy endpoint 2: mean Change in Time in Range (TIR) | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 2: mean Change in Time in Range
Efficacy endpoint 3: In patients with baseline abnormal Alanine Transaminase (ALT), Aspartate Aminotransferase (AST), and Gamma Glutamyl Transferase (GGT) values, change in ALT, AST, GGT | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 3: In patients with baseline abnormal ALT, AST and GGT values, change in ALT, AST, GGT
Efficacy endpoint 4: Change in body weight | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 4: Change in body weight
Efficacy endpoint 5: Change in Fasting C-peptide | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 5: Change in Fasting C-peptide
Efficacy endpoint 6: Change in FPG | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 6: Change in FPG
Efficacy endpoint 7: Change in homeostasis model assessment for insulin resistance (HOMA-IR) | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 7: Change in HOMA-IR
Efficacy endpoint 8: Change in Framingham Risk Score-Cardiovascular risk score (FRS-CVD) | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 8: Change in Framingham Risk Score-Cardiovascular risk score (FRS-CVD)
Efficacy endpoint 9: Change in MRI-proton density fat fraction (MRI-PDFF) | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 9: Change in MRI-PDFF
Efficacy endpoint 10: Achievement of HbA1c ≤ 53 mmol/mol (7.0%) | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 10: Achievement of HbA1c ≤ 53 mmol/mol (7.0%)
Efficacy endpoint 11: Change in food intake (amount of calories, fat, carbohydrates, proteins etc.) based on intake registration data | Through study completion, an average of 1 or 1,5 years
  Efficacy endpoint 11: Change in food intake (amount of calories, fat, carbohydrates, proteins etc.) based on intake registration data
Mechanistic: Change in resection tissue findings in morphological features | Week 12 after (re)DMR
  Mechanistic: Change in morphological features
Mechanistic: Change in resection tissue findings in functional level changes | Week 12 after (re)DMR
  Mechanistic: Change in functional level changes
Mechanistic: Change in resection tissue findings in cellular level changes | Week 12 after (re)DMR
  Mechanistic: Change in cellular level changes
Mechanistic: Mean Changes in small intestinal biopsy gene expression | Week 12 after (re)DMR
  Mechanistic: Mean Changes in small intestinal biopsy gene expression
Mechanistic: Mean Changes in small intestinal biopsy metabolomics/proteomics | Week 12 after (re)DMR
  Mechanistic: Mean Changes in small intestinal biopsy metabolomics /proteomics
Mechanistic: Change in Plasma Citrulline | Through study completion, an average of 1 or 1,5 years
  Mechanistic: Change in Plasma Citrulline
Mechanistic: Change in Cystatin Value | Through study completion, an average of 1 or 1,5 years
  Mechanistic: Change in Cystatin Value

CONTACTS AND LOCATIONS:
Overall Officials: Jacques JG Bergman, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam UMC, locatie VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for people that are interested in participating. — https://onderzoekdiabetes.nl/